CLINICAL TRIAL: NCT01466387
Title: A Phase 3b, Randomized, Open-Label Study to Evaluate the Safety and Immunogenicity of Select Travel Vaccines When Administered Concomitantly With Novartis Meningococcal ACWY Conjugate Vaccine in Healthy Adults
Brief Title: A Phase 3b, Randomized, Open-Label Study to Evaluate the Safety and Immunogenicity of Select Travel Vaccines When Administered Concomitantly With MenACWY in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59_38; 2011-000475-14 (EudraCT Number)
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis; Typhoid; Yellow Fever; Rabies; Japanese Encephalitis
Keywords: Adults; international travel vaccination; Meningococcal disease; meningococcal meningitis; typhoid; yellow fever; rabies; Japanese encephalitis
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Typhoid Fever; Yellow Fever; Rabies; Encephalitis, Japanese | interventions — Vi polysaccharide vaccine, typhoid; Yellow Fever Vaccine; Japanese Encephalitis Vaccines; Rabies Vaccines; MenACWY-CRM vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- TF+YF (Active Comparator): Subjects ≥18 years to ≤60 years of age who received one dose of typhoid Vi polysaccharide and yellow fever vaccine.
  Interventions: Biological: Typhoid Vi Polysaccharide Vaccine; Biological: Yellow Fever Vaccine
- TF + YF + MenACWY-CRM197 (Active Comparator): Subjects ≥18 years to ≤60 years of age who received one dose of typhoid Vi polysaccharide, yellow fever and meningococcal ACWY conjugate vaccine.
  Interventions: Biological: Typhoid Vi Polysaccharide Vaccine; Biological: Yellow Fever Vaccine; Biological: MenACWY-CRM Vaccine
- JE + Rabies (Active Comparator): Subjects ≥18 years to ≤60 years of age who received two doses of Japanese encephalitis and three doses of Rabies vaccine.
  Interventions: Biological: Japanese Encephalitis Vaccine; Biological: Rabies Vaccine
- JE + Rab + MenACWY-CRM197 (Active Comparator): Subjects ≥18 years to ≤60 years of age who received two doses of Japanese encephalitis and three doses of Rabies and one dose of meningococcal ACWY conjugate vaccine.
  Interventions: Biological: Japanese Encephalitis Vaccine; Biological: Rabies Vaccine; Biological: MenACWY-CRM Vaccine
- Rabies (Active Comparator): Subjects ≥18 years to ≤60 years of age who received three doses of Rabies vaccine.
  Interventions: Biological: Rabies Vaccine
- MenACWY-CRM197 (Combined) (Active Comparator): Subjects ≥18 years to ≤60 years of age who received one dose of meningococcal ACWY conjugate vaccine.
  Interventions: Biological: MenACWY-CRM Vaccine

INTERVENTIONS:
Biological: Typhoid Vi Polysaccharide Vaccine — One dose of typhoid Vi polysaccharide vaccine.
  Arms: TF + YF + MenACWY-CRM197; TF+YF
Biological: Yellow Fever Vaccine — One dose of yellow fever vaccine.
  Arms: TF + YF + MenACWY-CRM197; TF+YF
Biological: Japanese Encephalitis Vaccine — Two doses of Japanese Encephalitis Vaccine.
  Arms: JE + Rab + MenACWY-CRM197; JE + Rabies
Biological: Rabies Vaccine — Three doses of Rabies vaccine.
  Arms: JE + Rab + MenACWY-CRM197; JE + Rabies; Rabies
Biological: MenACWY-CRM Vaccine — One dose of MenACWY-CRM vaccine.
  Arms: JE + Rab + MenACWY-CRM197; MenACWY-CRM197 (Combined); TF + YF + MenACWY-CRM197

SUMMARY:
This study compares the safety and immunogenicity profile of several travel vaccines given alone or concomitantly with MenACWY-CRM to healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Female and male subjects who must be healthy and must be:

1. Between 18 and 60 years of age inclusive and who have given their written informed consent;
2. Available for all visits and telephone calls scheduled for the study;
3. In good health as determined by medical history, physical examination and clinical judgment of the investigator;
4. For female subjects, having a negative urine pregnancy test.

Exclusion Criteria:

Individuals not eligible to be enrolled in the study are those:

1. who are breastfeeding;
2. who have a personal history of Neisseria meningitidis infection, typhoid fever, rabies, or any flavivirus infection (e.g., Japanese encephalitis, tick-borne encephalitis, yellow fever, dengue fever, West Nile virus infection);
3. who have been immunized with any of the study vaccines within the last five years as determined by medical history and/or vaccination card;
4. who have received investigational agents or vaccines within 30 days prior to enrollment or who expect to receive an investigational agent or vaccine prior to completion of the study;
5. who have received live licensed vaccines within 30 days and inactive vaccine within 15 days prior to enrollment or for whom receipt of a licensed vaccine is anticipated during the study period.

   (Exception: Influenza vaccine may be administered up to 15 days prior to each study immunization and no less than 15 days after each study immunization);
6. who have received an anti-malaria drug, up to 2 months prior to the study;
7. who have experienced, within the 7 days prior to enrollment, significant acute infection (for example requiring systemic antibiotic treatment or antiviral therapy) or have experienced fever (defined as body temperature ≥ 38°C) within 3 days prior to enrollment;
8. who have any serious acute, chronic or progressive disease such as:

   * history of cancer
   * complicated diabetes mellitus
   * advanced arteriosclerotic disease
   * autoimmune disease
   * HIV infection or AIDS
   * blood dyscrasias
   * congestive heart failure
   * renal failure
   * severe malnutrition (Note: Subjects with mild asthma are eligible for enrollment. Subjects with moderate or severe asthma requiring routine use of inhaled or systemic corticosteroids are not eligible for enrollment);
9. who have epilepsy, any progressive neurological disease or history of Guillain-Barre syndrome;
10. who have a history of anaphylaxis, serious vaccine reactions, or allergy to any vaccine component, including but not limited to latex allergy, egg allergy, antibiotic allergy, chicken proteins or gelatin allergy;
11. who have a known or suspected impairment/alteration of immune function, either congenital or acquired or resulting from (for example):

    * receipt of immunosuppressive therapy within 30 days prior to enrollment (systemic corticosteroids administered for more than 5 days, or in a daily dose > 1 mg/kg/day prednisone or equivalent during any of 30 days prior to enrollment, or cancer chemotherapy);
    * receipt of immunostimulants;
    * receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 90 days prior to enrollment and for the full length of the study;
12. who are known to have a bleeding diathesis, or any condition that may be associated with a prolonged bleeding time;
13. who have myasthenia gravis; thyroid or thymic disorders,
14. who have any condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives;
15. who are part of the study personnel or close family members of those conducting this study.
16. for whom a long-term stay (≥ 1 month) was planned in Africa, Latin America, or Asia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 552 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Centrum ockovani a cestovni mediciny (Vaccination and Travel Medicine Centre) Poliklinika II, Bratri Stefanu 895, Hradec Kralove, Czechia
- Germany (4):
  - Bernhard Nocht Strasse 74, Hamburg
  - Berliner Centrum Fur Reise und Tropenmedizin, Jaegerstrasse 67-69, State of Berlin
  - University of Munich Georgenstr.5, München
  - Universitat Rostock, Ernst Heydemann Str 6, Rostock

REFERENCES:
- [Derived] Alberer M, Burchard G, Jelinek T, Reisinger E, Beran J, Hlavata LC, Forleo-Neto E, Dagnew AF, Arora AK. Safety and immunogenicity of typhoid fever and yellow fever vaccines when administered concomitantly with quadrivalent meningococcal ACWY glycoconjugate vaccine in healthy adults. J Travel Med. 2015 Jan-Feb;22(1):48-56. doi: 10.1111/jtm.12164. Epub 2014 Oct 13. PMID 25308927
- [Derived] Alberer M, Burchard G, Jelinek T, Reisinger E, Beran J, Meyer S, Forleo-Neto E, Gniel D, Dagnew AF, Arora AK. Co-administration of a meningococcal glycoconjugate ACWY vaccine with travel vaccines: a randomized, open-label, multi-center study. Travel Med Infect Dis. 2014 Sep-Oct;12(5):485-93. doi: 10.1016/j.tmaid.2014.04.011. Epub 2014 May 9. PMID 24873986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 5 sites (Berhard Nocht Institut, Germany, Berliner Centrum fuer Reise, Germany, Universitat Rostock, Germany, University of Munich, Germany, Vacc and Travel Med. Center, Czech Republic)
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- TF+YF+MenACWY-CRM197: Subjects ≥18 years to ≤60 years of age who received one dose of typhoid Vi polysaccharide, yellow fever and meningococcal ACWY conjugate vaccine.
- JE+Rabies: Subjects ≥18 years to ≤60 years of age who received two doses of Japanese encephalitis and three doses of Rabies vaccine.
- JE+Rabies+MenACWY-CRM197: Subjects ≥18 years to ≤60 years of age who received two doses of Japanese encephalitis and three doses of Rabies and one dose of meningococcal ACWY conjugate vaccine.
Period: Overall Study
Arm/Group | TF+YF | TF+YF+MenACWY-CRM197 | JE+Rabies | JE+Rabies+MenACWY-CRM197 | Rabies | MenACWY-CRM197 (Combined)
Started | 101 | 100 | 99 | 101 | 51 | 100
Completed | 100 | 100 | 98 | 99 | 51 | 99
Not Completed | 1 | 0 | 1 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TF+YF | TF+YF+MenACWY-CRM197 | JE+Rabies | JE+Rabies+MenACWY-CRM197 | Rabies | MenACWY-CRM197 (Combined) | Total
Number analyzed (Participants) | 101 | 100 | 99 | 101 | 51 | 100 | 552
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (10.8) | 35.1 (11.0) | 35.0 (11.5) | 35.0 (11.1) | 35.8 (11.6) | 36.9 (11.2) | 35.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 44 | 53 | 50 | 21 | 50 | 267
  Male | 52 | 56 | 46 | 51 | 30 | 50 | 285

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Anti-typhoid Vi Antibody Concentrations
Description: Assessment was made to demonstrate the non-inferiority of the geometric mean anti-typhoid Vi antibody concentrations, 28 days after the vaccination of typhoid Vi polysaccharide (TF) and yellow fever (YF) vaccines given concomitantly with MenACWY-CRM197 to typhoid Vi polysaccharide and yellow fever vaccines given alone in healthy adults aged ≥18 years to ≤60 years.
Time Frame: Baseline and 1 month postvaccination (day 29).
Population: Analysis was done on the per-protocol (PP) set, ie, the subjects who received the vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violations as defined prior to analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: El.U/mL
Arm/Group | TF+YF | TF+YF+MenACWY-CRM197
Number analyzed (Participants) | 100 | 99
El.U/mL
  Day 1 (Typhoid Fever) | 6.37 [5.3 to 7.65] | 5.6 [4.66 to 6.73]
  Day 29 (Typhoid Fever) | 134 [104 to 174] | 153 [118 to 197]
Statistical Analysis 1: Comparison: TF+YF vs TF+YF+MenACWY-CRM197; The primary criterion for immunogenicity (postvaccination, day 29) was that the lower limit of the two-sided 95% confidence interval around the observed ratio of geometric mean concentrations between one dose of typhoid Vi polysaccharide and yellow fever vaccines given concomitantly with MenACWY-CRM197 to typhoid Vi polysaccharide and yellow fever vaccines given alone was greater than 0.5; Test type: Non-Inferiority or Equivalence — GMC TF+YF+MenACWY-CRM/GMC TF+YF; ANCOVA — The testing was done by assessing the confidence interval of the ratio; The ANCOVA model included vaccine group and center as factors, age as covariate and was adjusted for baseline; Ratio of GMC = 1.14, 95% CI 2-sided [0.81 to 1.6]

2. Primary Outcome: Geometric Mean Anti-Yellow Fever Antibody Titer
Description: Assessment was made to demonstrate the non-inferiority of the geometric mean anti-yellow fever antibody titers, 28 days after the vaccination of typhoid Vi polysaccharide (TF) and yellow fever (YF) vaccines given concomitantly with MenACWY-CRM197 to typhoid Vi polysaccharide and yellow fever vaccines given alone in healthy adults aged ≥18 years to ≤60 years.
Time Frame: Baseline and 1 month postvaccination (day 29).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TF+YF | TF+YF+MenACWY-CRM197
Number analyzed (Participants) | 100 | 99
Titers
  Day 1 (Yellow Fever) | 9.05 [6.82 to 12] | 12 [8.68 to 15]
  Day 29 (Yellow Fever) | 5244 [3929 to 7000] | 5022 [3754 to 6717]
Statistical Analysis 1: Comparison: TF+YF vs TF+YF+MenACWY-CRM197; The primary criterion for immunogenicity (postvaccination, day 29) was that the lower limit of the two sided 95% CI around the observed ratio of geometric mean titers between one dose of typhoid Vi polysaccharide and yellow fever vaccines given concomitantly with MenACWY-CRM197 to typhoid Vi polysaccharide and yellow fever vaccines given alone was greater than 0.5; Test type: Non-Inferiority or Equivalence — GMT TF+YF+MenACWY/GMT TF+YF; ANCOVA — The testing was done by assessing the confidence interval of the ratio; The ANCOVA model included vaccine group and center as factors, age as covariate and was adjusted for baseline; Ratio of GMT. = 0.96, 95% CI 2-sided [0.65 to 1.41]

3. Primary Outcome: Geometric Mean Anti-Japanese Encephalitis Neutralizing Antibody Titers
Description: Assessment was made to demonstrate the non-inferiority of the geometric mean anti-Japanese encephalitis neutralizing antibody titers, 28 days after the vaccination of the second dose of Japanese Encephalitis vaccine and third dose of the rabies virus vaccine given concomitantly with MenACWY-CRM197 or alone in healthy adults aged ≥18 years to ≤60 years.
Time Frame: Baseline and 1 month post last vaccination (day 57).
Population: Analysis was done on the PP set, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violations as defined prior to analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- JE+Rab+MenACWY-CRM197: Subjects ≥18 years to ≤60 years of age who received two doses of Japanese Encephalitis and three doses of Rabies vaccine and one dose of Meningococcal conjugate vaccine.
Arm/Group | JE+Rabies | JE+Rab+MenACWY-CRM197
Number analyzed (Participants) | 96 | 97
Titers
  Day 1 (Japanese Encephalitis) | 5.61 [5.11 to 6.15] | 5.58 [5.09 to 6.12]
  Day 57 (Japanese Encephalitis) | 183 [151 to 221] | 165 [136 to 199]
Statistical Analysis 1: Comparison: JE+Rabies vs JE+Rab+MenACWY-CRM197; The primary criterion for immunogenicity (postvaccination, day 57) was that the lower limit of the two sided 95% CI around the observed ratio of geometric mean titers between the second dose of Japanese Encephalitis and third dose of rabies virus vaccines given concomitantly with MenACWY-CRM197 to Japanese Encephalitis and rabies virus vaccines given alone was greater than 0.5; Test type: Non-Inferiority or Equivalence — GMT JE + Rab + MenACWY-CRM/GMT JE + Rab; ANCOVA — The testing was done by assessing the confidence interval of the ratio; The ANCOVA model included vaccine group and centers as factors, age as covariate and was adjusted for baseline; Ratio of GMT = 0.9, 95% CI 2-sided [0.7 to 1.16]

4. Primary Outcome: Geometric Mean Anti-Rabies Virus Neutralizing Antibody Concentration
Description: Assessment was made to demonstrate the non-inferiority of the geometric mean anti-rabies virus neutralizing antibody concentrations, 28 days after the vaccination of the second dose of Japanese encephalitis vaccine and third dose of rabies virus vaccine given concomitantly with MenACWY-CRM197 or alone in healthy adults aged ≥18 years to ≤60 years.
Time Frame: Baseline and 1 month post last vaccination (day 57).
Population: Analysis was done on the per-protocol (PP) set, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violations as defined prior to analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | JE+Rabies | JE+Rab+MenACWY-CRM197
Number analyzed (Participants) | 96 | 97
IU/mL
  Day 1 (Rabies) | 0.056 [0.05 to 0.062] | 0.049 [0.044 to 0.054]
  Day 57 (Rabies) | 12 [9.68 to 14] | 11 [8.84 to 13]
Statistical Analysis 1: Comparison: JE+Rabies vs JE+Rab+MenACWY-CRM197; The primary criterion for immunogenicity (postvaccination, day 57) was that the lower limit of the two sided 95% CI around the observed ratio of geometric mean concentrations between the second dose of Japanese encephalitis and third dose of rabies virus vaccines given concomitantly with MenACWY-CRM197 to Japanese encephalitis and rabies virus vaccines given alone was greater than 0.5; Test type: Non-Inferiority or Equivalence — GMC JE + Rab + MenACWY-CRM/GMC JE + Rab; ANCOVA — The testing was done by assessing the confidence interval of the ratio; The ANCOVA model included vaccine group and center as factors, age as covariate and was adjusted for baseline; Ratio of GMC = 0.91, 95% CI 2-sided [0.71 to 1.17]

5. Secondary Outcome: Percentages Of Subjects With Anti-YF Neutralizing Antibody Titers ≥ 1/10, 28 Days After The Vaccination Of Typhoid Vi Polysaccharide And Yellow Fever, Concomitantly With MenACWY-CRM197 Or Given Alone
Description: Immunogenicity was assessed as the percentages of subjects who achieved seroprotection as measured by neutralization test for anti-YF neutralizing antibody titers after the vaccination of typhoid Vi polysaccharide and yellow fever, given alone or concomitantly with MenACWY-CRM197 on day 29.
  Seroprotection is defined as percentages of subjects who achieved anti-YF neutralizing antibody titers ≥ 1/10 on day 29.
Time Frame: Baseline and 1 month postvaccination (day 29).
Population: Analysis was done on the Modified-Intention to Treat (MITT) set, i.e. the subjects who provided evaluable serum samples whose assay results are available for at least one antigen on baseline and on at least one post-baseline visit.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TF+YF | TF+YF+MenACWY-CRM197
Number analyzed (Participants) | 100 | 100
Percentages of subjects
  Day 1 (Yellow Fever) | 34 [25 to 44] | 36 [27 to 46]
  Day 29 (Yellow Fever) | 100 [96 to 100] | 97 [91 to 99]

6. Secondary Outcome: Percentages Of Subjects With Anti-JE Neutralizing Antibody Titers ≥ 1/10, 28 Days After The Vaccination Of The Last Doses Of Japanese Encephalitis And Rabies, Given Concomitantly With MenACWY-CRM197 Or Alone
Description: Immunogenicity was measured as the percentages of subjects who achieved seroprotection as measured by neutralization test for anti-Japanese encephalitis neutralizing antibody titers, 28 days after administration of the second dose of Japanese encephalitis virus vaccine and 28 days after the vaccination of third dose of rabies virus vaccine, given alone or concomitantly with MenACWY-CRM197.
  Seroprotection is defined as percentages of subjects who achieved anti-JE neutralizing titers ≥ 1/10 on Day 57.
Time Frame: Baseline and 1 month post last vaccination (day 57).
Population: The analysis was done on the MITT data set.
Measure: Number (95% Confidence Interval); unit: Percentages of subects
Arm/Group | JE+Rabies | JE+Rabies+MenACWY-CRM197
Number analyzed (Participants) | 98 | 99
Percentages of subects
  Day 1 (Japanese Encephalitis) | 3 [1 to 9] | 4 [1 to 10]
  Day 57 (Japanese Encephalitis) | 99 [94 to 100] | 98 [93 to 100]

7. Secondary Outcome: Percentages Of Subjects With Anti-Rabies Virus Antibody Concentrations ≥ 0.5 IU/mL 28 Days After the Vaccination Of The Last Doses Of Japanese Encephalitis And Rabies Virus, Given Concomitantly With MenACWY-CRM197 Or Alone
Description: Immunogenicity was assessed as the percentages of subjects who achieved seroprotection as measured by neutralization test for anti-rabies neutralizing antibody titers, 28 days after administration of the second dose of Japanese encephalitis virus vaccine and 28 days after the vaccination of third dose of rabies virus vaccine, given alone or concomitantly with MenACWY-CRM197.
  Seroprotection is defined as a subject with a baseline hSBA titer < 1:4, seroresponse was defined as a post-vaccination hSBA titer ≥ 1:8; for a subject with a baseline hSBA titer ≥ 1:4, seroresponse was defined as a post-vaccination hSBA titer of at least 4 times the baseline.
Time Frame: Baseline and 1 month post last vaccination (day 57).
Population: Analysis was done on the MITT data set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- JE+Rabies+MenACWY-CRM197: Subjects ≥18 years to ≤60 years of age who received two doses of Japanese Encephalitis and three doses of Rabies vaccine and one dose of Meningococcal conjugate vaccine.
Arm/Group | JE+Rabies | JE+Rabies+MenACWY-CRM197
Number analyzed (Participants) | 98 | 99
Percentages of subjects
  Day 1 (Rabies) | 3 [1 to 9] | 1 [0.026 to 5]
  Day 57 (Rabies) | 100 [96 to 100] | 100 [96 to 100]

8. Secondary Outcome: Geometric Mean hSBA Titers For Meningococcal Serogroups A,C,W,Y 28 Days After The Vaccination Of MenACWY-CRM197 Given Concomitantly With Typhoid Vi Polysaccharide And Yellow Fever Vaccines Alone
Description: Immunogenicity was assessed by Serum Bactericidal Assay using human complement (hSBA) geometric mean titers (GMTs) for meningococcal serogroups A,C,W,Y 28 days after administration of MenACWY-CRM197 given concomitantly with typhoid Vi polysaccharide and yellow fever vaccines or alone.
Time Frame: Baseline and 1 month postvaccination (day 29).
Population: Analysis was done on the MITT data set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-CRM197 (Combined) | TF+YF+MenACWY-CRM197
Number analyzed (Participants) | 99 | 100
titers
  Serogroup A (Day 1) | 2.94 [2.43 to 3.56] | 2.78 [2.3 to 3.36]
  Serogroup A (Day 29) | 65 [44 to 95] | 62 [42 to 90]
  Serogroup C (Day 1) | 7.94 [5.94 to 11] | 7.03 [5.27 to 9.38]
  Serogroup C (Day 29) | 49 [35 to 70] | 54 [38 to 76]
  Serogroup W (Day 1) | 50 [35 to 71] | 32 [22 to 45]
  Serogroup W (Day 29) | 129 [94 to 177] | 211 [154 to 290]
  Serogroup Y (Day 1) | 7.61 [5.71 to 10] | 7.76 [5.83 to 10]
  Serogroup Y (Day 29) | 89 [62 to 129] | 78 [54 to 113]

9. Secondary Outcome: Seroresponse Rate For Meningococcal Serogroups A,C,W,Y 28 Days After Vaccination of MenACWY-CRM197 Given Concomitantly With Typhoid Vi Polysaccharide and Yellow Fever Vaccines or Alone
Description: Immunogenicity was assessed by seroresponse rates as measured by human serum bactericidal activity (hSBA) titers for meningococcal serogroups A,C,W,Y 28 days after administration of MenACWY-CRM197 given concomitantly with typhoid Vi polysaccharide and yellow fever vaccines or alone.
  Seroresponse is defined as a postvaccination hSBA titer ≥1:8; for a subject with a baseline hSBA titer ≥1:4, seroresponse is defined as a postvaccination hSBA titer of at least four times the baseline.
Time Frame: 1 month postvaccination (day 29)
Population: The analysis was done on the MITT data set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TF + YF + MenACWY-CRM197 | MenACWY-CRM197 (Combined)
Number analyzed (Participants) | 100 | 99
Percentages of subjects
  Serogroup A (Overall Seroresponse) | 72 [62 to 81] | 71 [61 to 79]
  Serogroup C (Overall Seroresponse) | 48 [38 to 58] | 47 [37 to 58]
  Serogroup W (Overall Seroresponse) | 51 [40 to 61] | 30 [21 to 40]
  Serogroup Y (Overall Seroresponse) | 63 [53 to 72] | 66 [55 to 75]

10. Secondary Outcome: Geometric Mean hSBA Titers for Meningococcal Serogroups A,C,W,Y 28 Days After the Vaccination of MenACWY-CRM197 Given Concomitantly With Japanese Encephalitis and Rabies Virus Vaccines or Alone
Description: Immunogenicity was measured by human serum bactericidal activity (hSBA) geometric mean titers (GMTs) for meningococcal serogroups A,C,W,Y 28 days after administration of MenACWY-CRM197 given concomitantly with Japanese encephalitis and rabies virus vaccines or alone.
Time Frame: Baseline and 1 month post last vaccination (day 29 or day 57).
Population: The analysis was done on the MITT data set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | JE + Rab + MenACWY-CRM197 | MenACWY-CRM197 (Combined)
Number analyzed (Participants) | 99 | 99
titers
  Serogroup A (Day 1) | 3.21 [2.65 to 3.88] | 2.94 [2.43 to 3.56]
  Serogroup A (Day 29 or Day 57) | 32 [22 to 47] | 65 [44 to 95]
  Serogroup C (Day 1) | 8.81 [6.59 to 12] | 7.94 [5.94 to 11]
  Serogroup C (Day 29 or Day 57) | 44 [31 to 62] | 49 [35 to 70]
  Serogroup W (Day 1) | 54 [38 to 77] | 50 [35 to 71]
  Serogroup W (Day 29 or Day 57) | 119 [87 to 164] | 129 [94 to 177]
  Serogroup Y (Day 1) | 8.11 [6.08 to 11] | 7.61 [5.71 to 10]
  Serogroup Y (Day 29 or Day 57) | 55 [38 to 80] | 89 [62 to 129]

11. Secondary Outcome: Seroresponse Rate for Meningococcal Serogroups A,C,W,Y 28 Days After Vaccination of MenACWY-CRM197 Given Concomitantly With Japanese Encephalitis and Rabies Virus Vaccines or Alone
Description: Immunogenicity was assessed by seroresponse rates as measured by human serum bactericidal activity (hSBA) titers for meningococcal serogroups A,C,W,Y 28 days after administration of MenACWY-CRM197 given concomitantly with Japanese encephalitis and rabies virus vaccines or alone.
  Seroresponse is defined as a subject with a baseline hSBA titer < 1:4, seroresponse was defined as a post-vaccination hSBA titer ≥ 1:8; for a subject with a baseline hSBA titer ≥ 1:4, seroresponse was defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 1 month post last vaccination (day 29 or day 57)
Population: The analysis was done on the MITT data set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | JE + Rab + MenACWY-CRM197 | MenACWY-CRM197 (Combined)
Number analyzed (Participants) | 99 | 99
Percentages of subjects
  Serogroup A (Overall Seroresponse) | 60 [49 to 69] | 71 [61 to 79]
  Serogroup C (Overall Seroresponse) | 43 [33 to 54] | 47 [37 to 58]
  Serogroup W (Overall Seroresponse) | 32 [23 to 42] | 30 [21 to 40]
  Serogroup Y (Overall Seroresponse) | 56 [45 to 66] | 66 [55 to 75]

12. Secondary Outcome: Geometric Mean Rabies Virus Neutralizing Antibody Concentration 28 Days After the Last Vaccination Of Rabies Virus Vaccine Concomitantly Either With Japanese Encephalitis or With Japanese Encephalitis And MenACWY-CRM197
Description: The immunogenicity was assessed in rabies virus vaccine as measured by geometric mean rabies virus neutralizing antibody concentration, 28 days after vaccination of the third dose, when administered alone or concomitantly either with Japanese encephalitis vaccine or with Japanese Encephalitis and MenACWY-CRM197 vaccines.
Time Frame: Baseline and 1 month post last vaccination (day 57).
Population: The analysis was done on the MITT data set.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- JE + Rabies + MenACWY-CRM197: Subjects ≥18 years to ≤60 years of age who received two doses of Japanese Encephalitis and three doses of Rabies and one dose of meningococcal ACWY conjugate vaccine.
Arm/Group | JE + Rabies + MenACWY-CRM197 | JE + Rabies | Rabies
Number analyzed (Participants) | 99 | 98 | 51
IU/mL
  Day 1 (Rabies) | 0.051 [0.044 to 0.059] | 0.057 [0.049 to 0.065] | 0.068 [0.056 to 0.082]
  Day 57 (Rabies) | 11 [8.84 to 13] | 11 [9.49 to 14] | 8.97 [6.98 to 12]

13. Secondary Outcome: Percentages of Subjects With Anti-rabies Virus Concentrations ≥ 0.5 IU/mL, 28 Days After the Last Vaccination of Rabies Virus Vaccine Concomitantly Either With Japanese Encephalitis or With Japanese Encephalitis and MenACWY-CRM197
Description: Immunogenicity was measured as the percentages of subjects who achieved seroprotection of anti-rabies virus antibody concentrations 28 days after vaccination of the third dose of rabies virus vaccine, when administered alone or concomitantly either with Japanese encephalitis or with Japanese encephalitis and MenACWY-CRM197 vaccines.
  Seroprotection is defined as percentages of subjects who achieved anti-rabies virus antibody concentrations ≥ 0.5 IU/mL on day 57.
Time Frame: Baseline and 1 month post last vaccination (day 57).
Population: The analysis was done on the MITT data set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- Rabies: Subjects ≥18 years to ≤60 yars of age who received three doses of Rabies vaccine.
Arm/Group | JE + Rabies + MenACWY-CRM197 | JE + Rabies | Rabies
Number analyzed (Participants) | 99 | 98 | 51
Percentages of subjects
  Day 1 (Rabies) | 1 [0.026 to 5] | 3 [1 to 9] | 8 [2 to 19]
  Day 57 (Rabies) | 100 [96 to 100] | 100 [96 to 100] | 100 [93 to 100]

14. Secondary Outcome: Number of Subjects With Adverse Events of Special Interest After Any Vaccination of Japanese Encephalitis and Rabies Virus Vaccines Given Concomitantly With MenACWY-CRM197 or Alone
Description: In addition to the AEs and SAEs. Additional AESI were collected from day 1 to day 57 postvaccination in subjects after the vaccination of Japanese encephalitis and rabies virus vaccines given concomitantly with MenACWY-CRM197 or alone.
Time Frame: day 1 to day 57 post last vaccination
Population: Analysis was done on the safety data set, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: subjects
Arm/Group | JE + Rabies + MenACWY-CRM197 | JE + Rabies
Number analyzed (Participants) | 101 | 99
subjects
  Injection site erythema | 0 | 1
  Hypersensitivity | 1 | 0
  Paresthesia | 0 | 1
  Erythema | 1 | 0
  Pruritus | 1 | 1
  Hot flush | 1 | 0

ADVERSE EVENTS:
Time Frame: day 1 to day 29 (one month postvaccination); day 1 to day 57 (one month post last vaccination)
Description: AEs and SAEs were collected from day 1-29 for subjects vaccinated with typhoid Vi polysaccharide+YF +MenACWY-CRM197 or alone, from day 1-57 vaccinated with JE+rabies virus+MenACWY-CRM197 or alone and who received rabies vaccine alone.
Arm/Group | TF+YF | TF+YF+MenACWY-CRM197 | JE+Rabies | JE+Rabies+MenACWY-CRM197 | Rabies | MenACWY-CRM197 (Combined)
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/100 | 1/99 | 1/101 | 0/51 | 0/100
Other Adverse Events (participants affected / at risk) | 27/101 | 30/100 | 23/99 | 22/101 | 9/51 | 9/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TF+YF (N=101) | TF+YF+MenACWY-CRM197 (N=100) | JE+Rabies (N=99) | JE+Rabies+MenACWY-CRM197 (N=101) | Rabies (N=51) | MenACWY-CRM197 (Combined) (N=100)
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TF+YF (N=101) | TF+YF+MenACWY-CRM197 (N=100) | JE+Rabies (N=99) | JE+Rabies+MenACWY-CRM197 (N=101) | Rabies (N=51) | MenACWY-CRM197 (Combined) (N=100)
Injection site pain (General disorders) | 12 | 8 | 6 | 4 | 2 | 2
Headache (General disorders) | 7 | 10 | 9 | 5 | 5 | 4
Influenza like illness (General disorders) | 5 | 9 | 5 | 6 | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3 | 3 | 7 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No